CLINICAL TRIAL: NCT05690659
Title: Impact of Rehabilitative Ultrasonography Imaging on Core Muscles Function in Patients With Visceral Adiposity: Randomized Controlled Trail
Brief Title: Imaging on Core Muscles Function in Patients With Visceral Adiposity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deraya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: P.T.REC/012/003449
Record Dates: First submitted 2023-01-09; First posted 2023-01-19 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Obesity, Abdominal
MeSH Terms: conditions — Obesity, Abdominal | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cavitation ultrasonic lipolysis (Experimental): on abdomen 2 sesions / week for 10 sessions , Treatment head was griped perpendicular to abdomen, and make slow circular motion with marked pressure.2 sesions / week for 10 sessions
  Interventions: Other: device and exercise
- RUSI guided core muscle exercise (Experimental): 2 sesions / week for 10 sessions For diaphragm muscle the transducer was placed on the sub costal region to visualize diaphragm muscle on the screen aiming to use US as a visual feedback procedure. instructed to have 5 seconds to contract the diaphragm muscle by deep breathing and hold the contraction. At the end of the 5-second period, the image was saved on the screen, and the measurement of the resultant increase in thickness was performed. Each subject performed a total of 10 contractions (intervention session) For transverse abdominis exercise,. draw in your umbilicus toward the spine without moving back or pelvis, while comfortably breathing in and out," for 10 seconds hold and then 15 seconds rest in between, it was repeated 3 sets of ten while keeping the transducer perpendicular to the surface of the skin in a transverse plane halfway between the ASIS and the lower ribcage along the anterior axillary line
  Interventions: Other: device and exercise
- combination of cavitation and RUSI (Experimental): combination of cavitation and RUSI 2 sesions / week for 10 sessions
  Interventions: Other: device and exercise

INTERVENTIONS:
Other: device and exercise — cavitation ultrasonic device therapeutic exercise guided ultrasonography imaging

SUMMARY:
The purpose of this study is to determine the effect of cavitation ultrasonic lipolysis, RUSI guided core muscle exercise and their combination (cavitation ultrasonic lipolysis and RUSI guided core muscles exercise) on diaphragmatic excursion, transverse abdominis activation ratio, visceral fat thickness and waist circumference in patients with visceral adiposity patients with visceral adiposity will be recognized by nutrition specialist. 45 patients were distributed randomly into three groups. The first group will be treated with Cavitation lipolysis twice weekly. The second group was treated with rehabilitative ultrasound imaging (RUSI) guided core muscle exercise. The third group was treated with combination of cavitation and RUSI. patients will be examined with medical ultrasound imaging and tape measurement.

DETAILED DESCRIPTION:
- Inclusion criteria: Forty five subjects participated in this study. Age of participants ranged from 25 to 45 years. 3. Waist circumference was more than 102 cm for men and 88 cm for women 4. Body mass index (BMI) ranged from 25 to 29.9 (Kg / m2). 5. Subjects hadn't received drugs

Exclusion criteria:

1. history of spinal surgery or spinal fracture.
2. Serious diseases, such as heart disease, kidney, liver diseases, gastric ulcer or duodenal ulcer.
3. A history of bronchial asthma or any chest disease.
4. Uncontrolled diabetes or hypertension.
5. Patients with peacemaker or any metal implant on the treated area.
6. Cancer or patient with past history of tumor excision

ELIGIBILITY:
Inclusion Criteria:

* Forty five subjects participated in this study.
* Age of participants ranged from 25 to 45 years.
* Waist circumference was more than 102 cm for men and 88 cm for women
* Body mass index (BMI) ranged from 25 to 29.9 (Kg / m2).
* Subjects hadn't received drugs

Exclusion Criteria:

.history of spinal surgery or spinal fracture.

* Serious diseases, such as heart disease, kidney, liver diseases, gastric ulcer or duodenal ulcer.
* A history of bronchial asthma or any chest disease.
* Uncontrolled diabetes or hypertension.
* Patients with peacemaker or any metal implant on the treated area.
* Cancer or patient with past history of tumor excision.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
diaphragm excursion | five weeks
  by ultrasound imaging in centimeter
transverse abdominins contraction ratio | 5 weeks
  by ultrasound imaging in percent

SECONDARY OUTCOMES:
visceral fat thickness | 5 weeks
  by ultrasound imaging in centimeter
waist circumference | 5 weeks
  by tape measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Deraya university, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No